CLINICAL TRIAL: NCT02635217
Title: Same Day Bidirectional Endoscopies - Does the Sequence of Procedures or Choice of Insufflator Matter?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Queen's University (Other)
Responsible Party: Principal Investigator, Dr. Lawrence Hookey, Associate Professor, Medical Director Endoscopy Unit, Hotel Dieu Hospital, Queen's University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Bidirectional endoscopy study
Record Dates: First submitted 2015-12-14; First posted 2015-12-18 (Estimated); Last update posted 2018-05-09 (Actual); Status verified 2018-05

CONDITIONS: Anemia; Colon Polyps
Keywords: Colonoscopy; Esophagogastroduodenoscopy; Patient satisfaction; Bidirectional endoscopies
MeSH Terms: conditions — Anemia; Colonic Polyps; Patient Satisfaction | interventions — Endoscopy, Digestive System

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Group A1 (Experimental): EGD performed before the Colonoscopy with Carbon Dioxide insufflation.
  Interventions: Device: Carbon dioxide insufflation; Procedure: EGD (Esophagogastroduodenoscopy) before Colonoscopy
- Group A2 (Experimental): EGD performed before the Colonoscopy with room air insufflation.
  Interventions: Device: room air insufflation; Procedure: EGD (Esophagogastroduodenoscopy) before Colonoscopy
- Group B1 (Experimental): Colonoscopy performed before the EGD with Carbon Dioxide insufflation.
  Interventions: Device: Carbon dioxide insufflation; Procedure: Colonoscopy before EGD (Esophagogastroduodenoscopy)
- Group B2 (Experimental): Colonoscopy performed before the EGD with room air insufflation.
  Interventions: Device: room air insufflation; Procedure: Colonoscopy before EGD (Esophagogastroduodenoscopy)

INTERVENTIONS:
Device: Carbon dioxide insufflation — using an automated carbon dioxide insufflator the gas will be infused on demand during the endoscopies
  Arms: Group A1; Group B1
Device: room air insufflation — using standard care room air will be infused on demand
  Arms: Group A2; Group B2
Procedure: EGD (Esophagogastroduodenoscopy) before Colonoscopy — the order of endoscopies will be randomized as well
  Arms: Group A1; Group A2
Procedure: Colonoscopy before EGD (Esophagogastroduodenoscopy)
  Arms: Group B1; Group B2

SUMMARY:
Upper endoscopies (Esophagogastroduodenoscopies-EGDs) as well as a lower endoscopies (Colonoscopies) are routinely performed by gastroenterologists to assess the lining of patients' upper and lower gastrointestinal tracts using a video endoscope (a long tube with a video camera on the end). An EGD is performed to examine the upper digestive tract to look for areas of inflammation, ulcerations, or other abnormalities in the swallowing tube, stomach, or duodenal lining. Similarly, a colonoscopy is performed to directly visualize the large bowel for polyps, inflammation, or other abnormalities in the lower bowel lining.

During these procedures, room air is routinely used to insufflate (expand/inflate the stomach and the colon) to allow for better viewing of the lining of the upper and lower gastrointestinal tracts; however, recently the use of carbon dioxide (CO2) (instead of air) has been shown to possibly have less post-procedure patient discomfort. Additionally, when both procedures are performed in the same day, it is currently unknown as to which sequence of procedures is better overall -whether to perform the EGD before colonoscopy or vice versa.

The overall aim of our research is to compare patients' comfort, total amount of sedation used, and overall satisfaction with the procedures between four randomly allocated groups, to see which method of insufflation and which procedural sequence is better when both procedures need to be performed in the same day. We hypothesize that in patients requiring same day endoscopies, performing an EGD prior to Colonoscopy with carbon dioxide (CO2) used as an insufflator is the best tolerated sequence associated with decreased sedation use and increased patient satisfaction/comfort.

DETAILED DESCRIPTION:
Same day bi-directional endoscopies (EGD-esophagogastro-duodenoscopies and colonoscopies) are routinely performed in endoscopy units. Little however is known if the order of sequence of the two procedures (i.e. EGD (upper endoscopy) before colonoscopy (lower endoscopy) or vice-versa) is of any consequence. Those who favor performing EGDs prior to colonoscopies (EGD first approach) argue that the sedation necessary for EGD is then carried over to the colonoscopy and thus allows for a better tolerated colonoscopy. Additionally, abdominal bloating caused by insufflation of air during colonoscopy could lead to reduced tolerance of the subsequent EGD. Others however, argue that the gaseous distention of the small intestine caused by performing the EGD first leads to a more difficult and uncomfortable colonoscopy thereafter, likely due to a mechanical effect of air migrating to the proximal colon. Studies comparing procedural sequences in same day endoscopies have revealed conflicting results to date.

Some studies show that using the EGD first approach before allows for better procedural quality, decreased overall patient discomfort, less sedation, and a much higher chance of determining the diagnosis in the undifferentiated patient (e.g. occult GI bleeding). Other studies either show no difference in overall patient discomfort and satisfaction between both procedures, or even preference for colonoscopy before EGD. While some of these studies use moderate sedation, others use no sedation at all making generalization of these results difficult.

The use of carbon dioxide (CO2) for insufflation during upper and lower endoscopies has recently become popular over traditionally used room air, especially after studies revealed lesser post-procedure patient discomfort with the use of CO2. Whether its use affects the preferred sequence of procedures is still unknown.

Institutional variation across Canada regarding the sequence of procedures for same day bidirectional endoscopies is currently based on a combination of personal preferences and the few studies available. Given the absence of any formal guidelines in this area, we undertake the current study to test the hypothesis: In patients requiring same day bi-directional endoscopies, performing an EGD prior to Colonoscopy with carbon dioxide (CO2) used as an insufflator is the best tolerated sequence associated with decreased sedation use and increased patient satisfaction/comfort.

ELIGIBILITY:
Inclusion Criteria:

* any patient with a clinical indication for receiving same day bi-directional endoscopies.

Exclusion Criteria:

* prior bowel or gastrointestinal surgery(s) (exception: appendectomy, cholecystectomy, hernia repair)
* known obstructive or cancerous lesions,
* active inflammatory bowel disease,
* hereditary polyposis syndromes,
* allergies to fentanyl and/or midazolam (SOC endoscopy sedatives),
* difficulties with communication or conditions affecting ability to provide informed consent,
* neurologic conditions that affect breathing (e.g. GBS, ALS or myasthenia gravis),

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-01 (Actual); Primary Completion 2017-11 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
Overall patient satisfaction | Day 0 (post procedure)
  Validated patient questionnaires administered to patients after both procedures are complete (on Day 0) followed by a recall interview via phone (on Day 7 after the procedures).

SECONDARY OUTCOMES:
sedation use | day 0 (day of procedure)
  Total sedation calculated as a total cumulative dose administered.
patient comfort | day 0
  Patient comfort assessed by the nurses during the procedures using previously validated assessment scales.
Patient satisfaction | Day 7

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence Hookey, MD, Study Director — Queen's University
Locations (1):
- Hotel Dieu Hospital, Kingston, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cho JH, Kim JH, Lee YC, Song SY, Lee SK. Comparison of procedural sequences in same-day bidirectional endoscopy without benzodiazepine and propofol sedation: starting at the bottom or the top. J Gastroenterol Hepatol. 2010 May;25(5):899-904. doi: 10.1111/j.1440-1746.2009.06157.x. PMID 20546443
- [Background] Zuckerman G, Benitez J. A prospective study of bidirectional endoscopy (colonoscopy and upper endoscopy) in the evaluation of patients with occult gastrointestinal bleeding. Am J Gastroenterol. 1992 Jan;87(1):62-6. PMID 1728127
- [Background] Carter D, Lahat A, Papageorgiou NP, Goldstein S, Eliakim R, Bardan E. Comparison of procedural sequence in same-day consecutive bidirectional endoscopy using moderate sedation: a prospective randomized study. J Clin Gastroenterol. 2014 Mar;48(3):236-40. doi: 10.1097/MCG.0b013e3182a87e5f. PMID 24100751
- [Background] Choi JS, Youn YH, Lee SK, Choi JY, Kim HM, Kim YJ, Han KJ, Cho HG, Song SY, Cho JH. Which should go first during same-day upper and lower gastrointestinal endoscopy? A randomized prospective study focusing on colonoscopy performance. Surg Endosc. 2013 Jun;27(6):2209-15. doi: 10.1007/s00464-012-2741-2. Epub 2013 Jan 26. PMID 23355152
- [Background] Hsieh YH, Lin HJ, Tseng KC. Which should go first during same-day bidirectional endosocopy with propofol sedation? J Gastroenterol Hepatol. 2011 Oct;26(10):1559-64. doi: 10.1111/j.1440-1746.2011.06786.x. PMID 21615790
- [Background] Kavitha K, Bharathi R, et. al Same Day Dual Endoscopy: Does the Sequence Matter? Gastrointestinal Endoscopy (abstract) 63.5 (2006) AB 145.
- [Background] Sajid MS, Caswell J, Bhatti MI, Sains P, Baig MK, Miles WF. Carbon dioxide insufflation vs conventional air insufflation for colonoscopy: a systematic review and meta-analysis of published randomized controlled trials. Colorectal Dis. 2015 Feb;17(2):111-23. doi: 10.1111/codi.12837. PMID 25393051
- [Background] Kurien M, Din S, Dear KL, Elphick DA. Same day bidirectional endoscopy - does the procedural order matter? J Gastrointestin Liver Dis. 2012 Sep;21(3):328. No abstract available. PMID 23012681
- [Background] Rostom A, Ross ED, Dube C, Rutter MD, Lee T, Valori R, Bridges RJ, Pontifex D, Webbink V, Rees C, Brown C, Whetter DH, Kelsey SG, Hilsden RJ. Development and validation of a nurse-assessed patient comfort score for colonoscopy. Gastrointest Endosc. 2013 Feb;77(2):255-61. doi: 10.1016/j.gie.2012.10.003. PMID 23317691
- [Background] Munson GW, Van Norstrand MD, O'donnell JJ, Hammes NL, Francis DL. Intraprocedural evaluation of comfort for sedated outpatient upper endoscopy and colonoscopy: the La Crosse (WI) intra-endoscopy sedation comfort score. Gastroenterol Nurs. 2011 Jul-Aug;34(4):296-301. doi: 10.1097/SGA.0b013e3182248777. PMID 21814063
- [Background] Aronchick CA, Lipshutz WH, Wright SH, Dufrayne F, Bergman G. A novel tableted purgative for colonoscopic preparation: efficacy and safety comparisons with Colyte and Fleet Phospho-Soda. Gastrointest Endosc. 2000 Sep;52(3):346-52. doi: 10.1067/mge.2000.108480. PMID 10968848
- [Background] Rostom A, Jolicoeur E. Validation of a new scale for the assessment of bowel preparation quality. Gastrointest Endosc. 2004 Apr;59(4):482-6. doi: 10.1016/s0016-5107(03)02875-x. PMID 15044882